CLINICAL TRIAL: NCT06861322
Title: The Effects of Short Foot Exercises on Knee Muscle Tone, Knee Pain and Function, Balance, and Quality of Life in Patients with Flexible Flat Foot with Knee Pain
Brief Title: Effects of Short Foot Exercise on Knee Pain, Muscle Tone, Balance, and Quality of Life in Flexible Flatfoot Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, EUNGJOON LEE, Principal investigator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2025-01-016-003
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Flexible Flatfoot; Knee Pain; Balance Impairment; Quality of Life (QOL)
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short Foot Exercise + Conventional Physical Therapy (Experimental): Participants in this group will receive Short Foot Exercise (SFE) combined with Conventional Physical Therapy for four weeks.
  This intervention combination aims to determine whether Short Foot Exercise, in addition to conventional physical therapy, provides greater improvements in knee pain, muscle tone, balance, and quality of life compared to physical therapy alone.
  Interventions: Behavioral: Short Foot Exercise; Behavioral: Conventional Physical Therapy
- Conventional Physical Therapy (Active Comparator): Participants in this group will receive Conventional Physical Therapy only for four weeks.
  This control group serves as a baseline comparator, allowing researchers to assess whether adding Short Foot Exercise to conventional therapy provides additional benefits for knee pain, muscle function, balance, and quality of life.
  Interventions: Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Behavioral: Short Foot Exercise — * Description: Short Foot Exercise is a therapeutic exercise designed to strengthen intrinsic foot muscles and improve medial longitudinal arch stability.
  * Procedure: Participants will perform Short Foot Exercise twice daily, five times per week for four weeks. The exercise consists of progressive phases, starting with basic foot activation and advancing to resistance-based strengthening using bands.
  * Purpose: To determine if strengthening the foot's intrinsic muscles positively impacts knee pain, muscle function, and balance in individuals with flexible flatfoot.
  Arms: Short Foot Exercise + Conventional Physical Therapy
Behavioral: Conventional Physical Therapy — * Description: Standard non-invasive physical therapy aimed at reducing knee pain, improving muscle relaxation, and enhancing lower limb function.
  * Procedure: Participants will receive twice-weekly conventional physical therapy for ten minutes per session over four weeks. Treatment includes soft tissue mobilization, muscle relaxation techniques, and neuromuscular stimulation, as appropriate for knee pain relief.
  * Purpose: To evaluate its effectiveness as a standalone treatment compared to the addition of Short Foot Exercise.

SUMMARY:
This study was a clinical trial to investigate the effects of Short Foot Exercise (SFE) and standard physical therapy on knee muscle tone, knee pain and function, balance ability, and quality of life in adults with flexible flat feet and knee pain.

DETAILED DESCRIPTION:
This study aims to determine whether strengthening foot intrinsic muscles through SFE can reduce knee pain, improve muscle function, enhance balance, and improve quality of life in individuals with flexible flatfoot. Results may provide evidence-based rehabilitation strategies for managing knee pain in these patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index): If between 18 and 25 kg/m²
* Litigation period: If knee pain lasted for more than 6 weeks
* Navicular drop test: If it was 10 mm or more
* Numerical assessment scale: If knee pain was 4 or more
* Health status: If you are a person without health problems and are trying to participate in the experiment

Exclusion Criteria:

* History of knee surgery: If you have had knee surgery
* Treatment history: If you have received physical therapy for knee pain in the 4 weeks before the start of the study
* Mental status: If you have a psychological disorder that may interfere with your participation in the study
* Injury status: If you have a current serious injury affecting the lower extremity joints and foot
* Lower extremity alignment abnormalities and specific conditions: If you have structural flat foot, scoliosis
* Diseases and other conditions: If you have diabetes, rheumatoid arthritis, or menopause
* Neurological disorders: If you have experienced a neurological disorder within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-02 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Muscle Tension from Baseline to 4 Weeks (Measured by Myoton Pro - Frequency in Hz) | From enrollment to the end of treatment at 4 weeks
  * Description: This outcome measure assesses changes in muscle tension (tone) in the knee region before and after the intervention.
  * Measurement Tool: Myoton Pro
  * Unit of Measure: Frequency (Hz)
  * Assessment Method: Myoton Pro applies a gentle mechanical impulse to the skin overlying the Vastus Medialis, Biceps Femoris, Gastrocnemius Medialis, and Tibialis Anterior muscles, recording oscillation frequency as an indicator of muscle tone.
Change in Knee Muscle Stiffness from Baseline to 4 Weeks (Measured by Myoton Pro - Stiffness in N/m) | From enrollment to the end of treatment at 4 weeks
  * Description: This measure evaluates changes in muscle stiffness, reflecting muscle resistance to external force.
  * Measurement Tool: Myoton Pro
  * Unit of Measure: Newton per meter (N/m)
  * Assessment Method: Stiffness is quantified by Myoton Pro by applying a controlled impulse and measuring the muscle's resistance to deformation.
Change in Knee Muscle Elasticity from Baseline to 4 Weeks (Measured by Myoton Pro - Logarithmic Decrement) | From enrollment to the end of treatment at 4 weeks
  * Description: This measure evaluates changes in muscle elasticity, which indicates the muscle's ability to return to its original shape after deformation.
  * Measurement Tool: Myoton Pro
  * Unit of Measure: Logarithmic decrement
  * Assessment Method: The Myoton Pro records how quickly oscillations in the muscle dampen after a mechanical impulse, representing its elasticity.

SECONDARY OUTCOMES:
Change in Dynamic Balance from Baseline to 4 Weeks (Measured by Y-Balance Test - Reach Distance in cm) | From enrollment to the end of treatment at 4 weeks
  * Description: This measure assesses changes in lower limb balance and stability using the Y-Balance Test (YBT).
  * Measurement Tool: Y-Balance Test (YBT)
  * Unit of Measure: Reach distance (cm)
  * Assessment Method: Participants will perform three reach directions (anterior, posteromedial, posterolateral) while maintaining single-leg stance. The maximum reach distance for each direction is recorded and averaged.
Change in Quality of Life from Baseline to 4 Weeks (Measured by EQ-5D-5L - Score on a 5-Dimension Scale) | From enrollment to the end of treatment at 4 weeks
  * Description: This outcome measure evaluates self-reported quality of life in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  * Measurement Tool: EQ-5D-5L
  * Unit of Measure: Score on a 5-Dimension Scale
  * Assessment Method: Participants rate their health status on a 5-level Likert scale (1 = No problems, 5 = Extreme problems). A total EQ-5D-5L index score is calculated using a weighted algorithm.
Change in Knee Pain from Baseline to 4 Weeks (Measured by WOMAC Pain Subscale - Score on a 5-Point Likert Scale) | From enrollment to the end of treatment at 4 weeks
  * Description: This measure evaluates knee pain severity before and after treatment.
  * Measurement Tool: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Pain Subscale
  * Unit of Measure: Score on a 5-Point Likert Scale
  * Assessment Method: Participants rate pain intensity across five activities (e.g., walking, climbing stairs) using a 0-4 scale (0 = No pain, 4 = Extreme pain).
Change in Knee Function from Baseline to 4 Weeks (Measured by WOMAC Function Subscale - Score on a 5-Point Likert Scale) | From enrollment to the end of treatment at 4 weeks
  * Description: This measure assesses changes in functional ability and movement limitations.
  * Measurement Tool: WOMAC - Function Subscale
  * Unit of Measure: Score on a 5-Point Likert Scale
  * Assessment Method: Participants rate functional difficulty in 17 daily activities (e.g., rising from a chair, bending) on a 0-4 scale (0 = No difficulty, 4 = Extreme difficulty).

CONTACTS AND LOCATIONS:
Overall Officials: eungjoon lee, Study Director — Samyuk University
Locations (1):
- Samyuk University, Seoul, Nowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No